CLINICAL TRIAL: NCT01636297
Title: The Cyclical Lower-extremity Exercise for Parkinson's Trial
Acronym: CYCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Jay Alberts, Associate Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01NS073717-01 (NIH)
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Forced exercise (Experimental): Exercise on stationary cycle that was controlled by a motor to augment voluntary cycling rate by 35%
  Interventions: Behavioral: Forced exercise
- Voluntary Exercise (Experimental): Exercise on a stationary cycle without motor assistance
  Interventions: Behavioral: Voluntary exercise
- No Exercise (No Intervention): Participants received no exercise intervention and served as the control group

INTERVENTIONS:
Behavioral: Forced exercise — Exercise on a stationary cycle that was controlled by a motor, to augment voluntary cycling rate by 35%. Intervention was administered 3 times per week for 8 weeks
  Arms: Forced exercise
Behavioral: Voluntary exercise — Exercise on a stationary cycle without motor assistance. Intervention was administered 3 times per week for 8 weeks
  Arms: Voluntary Exercise

SUMMARY:
The purpose of this study is to gain a better understanding of how exercise training affects motor/hand function and brain function in those diagnosed with Parkinson's disease. The investigators want to study if exercise will improve hand function and improve the level of brain activity.

DETAILED DESCRIPTION:
Current medical and surgical approaches to Parkinson's disease (PD) are expensive and associated with a variety of side effects that may compromise the patient's quality of life. Development of a non-drug, non-surgical therapeutic approach to improve motor function would provide an attractive adjunct to current PD treatment approaches. Promising results from animal exercise studies have not been translated to patients with PD.

Animal studies suggest forced-exercise produces an endogenous increase in neurotrophic factors. An increase in these factors is believed to improve the capacity of dopamine neurons to deliver dopamine and selectively increase dopamine levels within the dorsolateral striatum. Models of PD provide a theoretical framework for forced-exercise and explain why voluntary exercise is not associated with global improvements in motor function for PD patients. Based on model predictions, decreased motor cortical activation limits PD patients' ability to perform voluntary exercise at the relatively high rate used in animal studies that demonstrate a therapeutic benefit. Therefore, PD patients may not be able to exercise (voluntarily) at sufficiently high rates to trigger the endogenous release of neurotrophic factors thought to underlie global improvements in motor functioning. A safe lower extremity forced-exercise paradigm that augments PD patients voluntary exercise rates has been developed for humans in an ongoing R21 project. Similar to our initial study, PD patients completing an 8-week forced-exercise intervention exhibited nearly a 25% percent improvement in clinical motor ratings, patients completing a voluntary exercise intervention showed no improvement in clinical ratings. Our recent fMRI data indicate that an acute bout of forced-exercise in PD patients produces a similar subcortical and cortical activation pattern as is seen following administration of levodopa. Global improvements in motor function and increased neural activity suggest forced-exercise may be altering brain function in PD patients. The goal of this project is to determine and compare the effects of forced versus voluntary exercise on PD motor and non-motor function and associated changes in the pattern of neural activity.

A single-center, parallel-group, rater-blind, study in a 2:2:1 randomization is proposed. A total of 100 mild to moderate idiopathic PD patients will be randomized to a voluntary, forced or no-exercise control group. Exercise groups will exercise at identical aerobic intensities, however those in the forced group will be provided mechanical assistance to perform exercise 35% faster than their voluntary exercise rate.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Clinical diagnosis of idiopathic PD. The diagnosis of PD will be based on the presence of at least two of the cardinal signs of this disorder (akine¬sia/bradykinesia, rest tremor, rigidity, gait and postural instability) with at least one of the signs being rest tremor or akinesia/bradykinesia.
* Hoehn and Yahr stage II-III when off PD medication.
* UPDRS motor score between 6-45 out of a maximum of 108 when off PD medication.
* Stable anti-parkinsonian medication for one month prior to study enrollment or consistent in desire to stay off anti-parkinson medication.
* Age between 30 and 75 years.

Exclusion Criteria:

* Clinically significant medical disease that would increase the risk of exercise-related complications (e.g. cardiac or pulmonary disease, diabetes mellitus, hypertension, stroke).
* Dementia as evidenced by a score less than 116 on the Mattis Dementia Rating Scale.
* Other medical or musculoskeletal contraindications to exercise.
* Undergone any surgical procedure for treatment of PD, DBS, pallidotomy or thalamotomy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Alberts, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Jansen AE, Koop MM, Rosenfeldt AB, Alberts JL. High intensity aerobic exercise improves bimanual coordination of grasping forces in Parkinson's disease. Parkinsonism Relat Disord. 2021 Jun;87:13-19. doi: 10.1016/j.parkreldis.2021.04.005. Epub 2021 Apr 20. PMID 33932704
- [Derived] Penko AL, Zimmerman NM, Crawford M, Linder SM, Alberts JL. Effect of Aerobic Exercise on Cardiopulmonary Responses and Predictors of Change in Individuals With Parkinson's Disease. Arch Phys Med Rehabil. 2021 May;102(5):925-931. doi: 10.1016/j.apmr.2020.12.011. Epub 2021 Jan 14. PMID 33453190
- [Derived] Rosenfeldt AB, Koop MM, Fernandez HH, Alberts JL. High intensity aerobic exercise improves information processing and motor performance in individuals with Parkinson's disease. Exp Brain Res. 2021 Mar;239(3):777-786. doi: 10.1007/s00221-020-06009-0. Epub 2021 Jan 4. PMID 33394100
- [Derived] Rosenfeldt AB, Rasanow M, Penko AL, Beall EB, Alberts JL. The cyclical lower extremity exercise for Parkinson's trial (CYCLE): methodology for a randomized controlled trial. BMC Neurol. 2015 Apr 24;15:63. doi: 10.1186/s12883-015-0313-5. PMID 25902768

RESULTS

PARTICIPANT FLOW:
Groups:
- Forced Exercise: Forced exercise: Exercise on a stationary cycle, controlled by motor , to augment voluntary rate by 35%
- Voluntary Exercise: Voluntary exercise: Exercise on a stationary bicycle without motor assistance
- No Exercise: No-exercise/control: No exercise intervention is given. This group serves as a control group.
Period: Overall Study
Arm/Group | Forced Exercise | Voluntary Exercise | No Exercise
Started | 40 | 40 | 20
Completed | 36 | 36 | 19
Not Completed | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Forced Exercise: Forced exercise: Exercise on a stationary bicycle, driven by a motor controlled by an algorithm, to force an individual to pedal faster than their voluntary cadence, 3 times per week for 8 weeks
- Voluntary Exercise: Voluntary exercise: Exercise on a stationary bicycle without augmenting cadence 3 times per week for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Forced Exercise | Voluntary Exercise | No Exercise | Total
Number analyzed (Participants) | 40 | 40 | 20 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8) | 61 (9) | 65 (6) | 63 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 6 | 42
  Male | 23 | 21 | 14 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 38 | 40 | 20 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 36 | 19 | 91

OUTCOME MEASURES:

1. Primary Outcome: MDS-UPDRS Motor III Score
Description: The Movement Disorder Society-Unified Parkinson's disease Rating Scale (MDS-UPDRS) Motor III Score is a subscale of the MDS-UPDRS. The MDS-UPDRS III is the sum of 33 scores that evaluate Parkinson's disease motor symptoms on a scale from 0 to 4 points. A score of 0 indicated no symptom is present and a maximum score of 4 indicates the most severe symptom, the total scale range is 0-132, where higher scores indicate more severe symptoms. The primary outcome is the change in total motor subscale score in the MDS-UPDRS from baseline versus the three end of treatment (EOT) assessments.
Time Frame: Change from baseline over 16 weeks
Measure: Mean (95% Confidence Interval); unit: change in MDS- UPDRS III score
Arm/Group | Forced Exercise | Voluntary Exercise | No Exercise
Number analyzed (Participants) | 36 | 36 | 19
change in MDS- UPDRS III score | -4.8 [-7.7 to -1.9] | -4.9 [-7.8 to -2.0] | 1.8 [-2.1 to 5.8]

2. Primary Outcome: Trail Making Test
Description: The Trail Making test is a test of executive function and the primary outcome is total test time. The total time that it takes to complete the test was recorded at baseline and then after the end of treatment. Test time recording begins with the start of the test and ends when the test is completed. Longer times indicate worse executive function. The outcome is the change in test time on the trail making test from baseline to the end of treatment (EOT) assessment.
Time Frame: Change from baseline over 16 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Forced Exercise | Voluntary Exercise | No Exercise
Number analyzed (Participants) | 35 | 34 | 19
seconds | -3.26 (4.49) | -2.91 (7.83) | -3.8 (3.36)

3. Primary Outcome: Number of Participants With Increased Motor Cortex and Thalamus Connectivity
Description: The primary outcome measure will number of patients that increased their connection between the motor cortex and the thalamus. The functional connection was assessed using functional magnetic resonance imaging. The outcome measure was change in connectivity from baseline to end of treatment.
Time Frame: Change from baseline to end of treatment
Population: A subgroup of participants from only the exercise groups were analyzed for this outcome measure, as not all participants in this study received functional MRI's. The No Exercise group was not included in this subgroup analysis and did not receive MRI.
Measure: Count of Participants; unit: Participants
Groups:
- Forced Exercise: Forced exercise: Exercise on a stationary cycle, controlled by a motor to augment voluntary rate by 35%
- Voluntary Exercise: Voluntary exercise: Exercise on a stationary cycle without motor assistance
Arm/Group | Forced Exercise | Voluntary Exercise | No Exercise
Number analyzed (Participants) | 6 | 6 | 0
Participants | 4 | 2 | 0

ADVERSE EVENTS:
Time Frame: Participants were enrolled for 16 weeks.
Groups:
- Forced Exercise: Forced exercise: Exercise on a stationary cycle that was controlled by a motor to augment voluntary rate by 35%
Arm/Group | Forced Exercise | Voluntary Exercise | No Exercise
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/19
Other Adverse Events (participants affected / at risk) | 1/36 | 0/36 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Forced Exercise (N=36) | Voluntary Exercise (N=36) | No Exercise (N=19)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No